CLINICAL TRIAL: NCT02014298
Title: LONG-TERM AND CONTINUED IMPROVEMENT OF MATURE BURN SCARS IN RESPONSE TO NONABLATIVE FRACTIONAL LASER - A RANDOMIZED CONTROLLED TRIAL WITH HISTOLOGICAL EVALUATION
Brief Title: Non Ablative Fractional Laser Treatment of Burn Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Taudorf, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H3-2009-149
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Burn Scars
Keywords: Burns; Non-ablative fractional laser; scar texture; histology; laser treatment; erbium:glass laser; meshed skin-grafts; photothermolysis; skin
MeSH Terms: conditions — Burns | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): One area assessed as a control area, compared to the laser-treated area
  Interventions: Radiation: non-ablative fractional laser
- Non-ablative Laser treatment (Active Comparator): 3 Non-ablative fractional laser treatments of one area
  Interventions: Other: control

INTERVENTIONS:
Radiation: non-ablative fractional laser — 3 treatments with 4-6 weeks interval
  Other Names: non-ablative fractional er:glass laser; 1,540 nm laser treatment
  Arms: Control
Other: control — observation, comparison to laser-treated area
  Other Names: observation
  Arms: Non-ablative Laser treatment

SUMMARY:
BACKGROUND: Increasing evidence appears for non-ablative fractional laser (NAFL) to remodel mature burn scars.

OBJECTIVES: To investigate long-term clinical and histological appearance of mature burn scars after NAFL-treatment.

HYPOTHESIS: That NAFL can modulate mature burn scars with subsequently improved cosmetic and functional appearance.

METHODS: Study patients with burn scars at trunk or extremities. Side-by-side test areas are randomized to three monthly 1,540 nm NAFL-treatments or control, followed by blinded evaluations at 1, 3, and 6 months using mPOSAS (modified Patient and Observer Scar Assessment Scale; 1 = normal skin, 10 = worst imaginable scar).

ELIGIBILITY:
Inclusion Criteria:

* legally competent adults aged 18-60 years
* Fitzpatrick skin type I-III
* burn scar 1 year or older
* total scar area allowing selection of two similar side-by-side test areas of minimum 1.5 × 3 cm for study purpose

Exclusion Criteria:

* pregnancy or lactation
* suntan
* wounds or infections in study area
* tendency to form hypertrophic scars or keloids
* oral retinoids, anti-inflammatory or immunosuppressive drugs within the last six months
* current anticoagulants
* previous treatments in test area with laser, Intense Pulsed Light, dermabrasion, chemical peel or filler.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in overall Scar-appearance | 1,3 and 6 months follow-up
  Primary endpoint is change in overall scar-appearance assessed by a slightly modified Patient and Observer Scar Assessment Scale (evaluation of study area omitted since this is fixed as part of study procedure). Scale: 1= normal skin; 10= worst imaginable scar.

SECONDARY OUTCOMES:
specific clinical and histological scar appearance | 1, 3, and 6 months follow-up
  Additional assessments include:
  * evaluation of vascularity, pigmentation, thickness, relief, pliability (evaluated on modified Patient and Observer Scar Assessment Scale)
  * histological changes (Small safety issue from taking a 4 mm cutaneous punch biopsy)
  * patient satisfaction
  * adverse events (pain during treatment, immediate treatment reaction, 24h treatment reaction, evaluation of side effects at 6 months follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, MD,PhD,DmSc, Study Director — Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Bispebjerg Hospital, University of Copenhagen, Copenhagen NV, Copenhagen, Denmark